CLINICAL TRIAL: NCT00024024
Title: A Phase I-II Trial Of BMS-275291 In Patients With HIV-Related Kaposi's Sarcoma
Brief Title: BMS-275291 in Treating Patients With HIV-Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02410; AMC-024; CPMC-IRB-13985; CDR0000068885 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-09-13; First posted 2003-08-05 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2008-04

CONDITIONS: Sarcoma
Keywords: AIDS-related Kaposi sarcoma; recurrent Kaposi sarcoma
MeSH Terms: conditions — Sarcoma; AIDS-related Kaposi sarcoma; Sarcoma, Kaposi | interventions — N-((2S)-2-mercapto-1-oxo-4-(3,4,4- trimethyl-2,5-dioxo-1-imidazolidinyl)butyl)-L-leucyl-N,3- dimethyl-L-Valinamide

ARMS (1):
- Arm I (Experimental): Patients receive oral BMS-275291 1-2 times daily. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 6 patients receive escalating doses of BMS-275291 until the recommended phase II dose (RPTD) is determined. The RPTD is the dose at which no more than 1 of 6 patients experiences dose-limiting toxicity and more than 1 of 6 patients experiences clinical response or at least 5 of 6 patients demonstrate biologic activity. An additional 29 patients are treated at the RPTD.
  Interventions: Drug: rebimastat

INTERVENTIONS:
Drug: rebimastat

SUMMARY:
Phase I/II trial to study the effectiveness of BMS-275291 in treating patients who have HIV-related Kaposi's sarcoma. Drugs such as BMS-275291 may stop the growth of Kaposi's sarcoma by stopping blood flow to the tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine whether the change in percent of apoptotic cells on tumor biopsies before and after treatment with BMS-275291 is a valid endpoint in patients with HIV-related Kaposi's sarcoma.

II. Determine the safety and tolerability of this drug in these patients. III. Determine the antitumor effects of this drug in these patients. IV. Determine the effect of this drug on overall quality of life and tumor-specific symptoms in these patients.

V. Determine the effect of this drug on CD4 and CD8 cell counts and percentages and HIV viral load in these patients.

VI. Determine the effect of this drug on human herpes virus-8 (HHV-8) viral load and correlate HHV-8 viral burden, tumor stage, and prognosis in these patients.

VII. Determine the peak plasma concentration of this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive oral BMS-275291 1-2 times daily. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients receive escalating doses of BMS-275291 until the recommended phase II dose (RPTD) is determined. The RPTD is the dose at which no more than 1 of 6 patients experiences dose-limiting toxicity and more than 1 of 6 patients experiences clinical response or at least 5 of 6 patients demonstrate biologic activity. An additional 29 patients are treated at the RPTD.

Quality of life is assessed on day 15 of the first course and then every 28 days thereafter.

Patients are followed for at least 1 month.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Kaposi's sarcoma (KS) with serologically documented HIV infection
* No symptomatic visceral KS requiring cytotoxic therapy unless refractory to or intolerant of all currently approved agents for visceral KS
* At least 5 measurable lesions

  * No prior local therapy to any indicator lesion unless clear progression has taken place since treatment

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count at least 750/mm3
* Platelet count at least 75,000/mm3
* Hemoglobin at least 8 g/dL

Hepatic:

* Bilirubin no greater than 1.0 times upper limit of normal (ULN) (no greater than 3.5 mg/dL if secondary to indinavir therapy provided direct bilirubin normal)
* AST and ALT no greater than 3 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance greater than 60 mL/min

Other:

* No acute, active opportunistic infection within the past 14 days except oral thrush or genital herpes
* No other serious medical illness within the past 14 days
* No other malignancy requiring cytotoxic therapy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior biologic therapy for KS and recovered

Chemotherapy:

* At least 3 weeks since prior chemotherapy for KS and recovered
* No concurrent systemic chemotherapy for KS

Endocrine therapy:

* No concurrent corticosteroids except replacement doses

Radiotherapy:

* At least 3 weeks since prior radiotherapy for KS and recovered

Other:

* All antiretroviral therapy must be at a stable dose for at least the past 4 weeks and during treatment
* At least 3 weeks since prior local therapy for KS and recovered
* At least 3 weeks since prior investigational therapy for KS and recovered
* At least 14 days since prior acute treatment of infections other than thrush and genital herpes
* Recovered from toxic effects of any other prior KS treatment
* No other concurrent investigational drugs except investigational new drug (IND)-available antiretroviral agents
* No other concurrent KS-specific treatment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2001-08; Primary Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Hayden Von Roenn, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (3):
- United States (3):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Herbert Irving Comprehensive Cancer Center, New York, New York

REFERENCES:
- [Result] Brinker BT, Krown SE, Lee JY, Cesarman E, Chadburn A, Kaplan LD, Henry DH, Von Roenn JH. Phase 1/2 trial of BMS-275291 in patients with human immunodeficiency virus-related Kaposi sarcoma: a multicenter trial of the AIDS Malignancy Consortium. Cancer. 2008 Mar 1;112(5):1083-8. doi: 10.1002/cncr.23108. PMID 18224669